CLINICAL TRIAL: NCT01230476
Title: Induction and Concurrent Chemoradiotherapy With Cetuximab for Patients With Locally Advanced Nasopharyngeal Carcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: University of Malaya (Other)
Collaborators: Merck Serono International SA (Industry)
Responsible Party: Principal Investigator, Ho Gwo Fuang, Medical Lecturer, University of Malaya
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EMR 62202-832
Record Dates: First submitted 2010-10-18; First posted 2010-10-29 (Estimated); Last update posted 2019-10-07 (Actual); Status verified 2019-10

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Locally advanced nasopharyngeal carcinoma; Neoadjuvant chemotherapy; Chemoradiation; Cetuximab
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cetuximab and chemotherapy (Experimental): 2 cycles of neoadjuvant cisplatin and 5FU (3 weekly), given with weekly cetuximab, followed by 7 doses of weekly cisplatin and cetuximab concurrent with radiotherapy
  Interventions: Drug: Cetuximab

INTERVENTIONS:
Drug: Cetuximab — Cetuximab loading dose of 400mg/m2, then weekly dose of 250mg/m2 for 12 doses; Neoadjuvant Cisplatin 75mg/m2 D1, 5FU 1000mg/m2 D2-5, for 2 cycles; Concurrent Cisplatin 30mg/m2 given with radiation 70Gy/35fraction/7weeks.

SUMMARY:
Standard of care for treatment of nasopharyngeal carcinoma is chemoradiation with concurrent cisplatin. Addition of a second agent, cetuximab, which targets nasopharyngeal carcinoma cells with high EGFR protein expression, may enhance the effectiveness of radiation and result in better tumour control. This study investigates the addition of 2 cycles of cisplatin/5FU chemotherapy with cetuximab, followed by cisplatin and cetuximab concurrent with radiation, for treatment of locally advanced nasopharyngeal carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* Inpatients or outpatients, 18-65 years of age
* Histologically confirmed, newly diagnosed locally advanced (UICC/AJCC stage III to IVB) nasopharyngeal carcinoma requiring radiotherapy
* Evidence of unidimensional measurable disease as per RECIST criteria
* No systemic metastatic disease (M0)
* ECOG performance status of 0 or 1 at study entry
* Effective contraception
* White blood cell count ≥ 3,000/mm3 with neutrophils ≥1,500/mm3, platelet count ≥100,000/mm3, hemoglobin ≥ 5.6 mmol/L (9 g/dL)
* Total bilirubin ≤ 1.5x upper reference range
* AST & ALT ≤ 1.5x upper reference range
* Glomerular filtration rate > 60 ml/min
* Serum creatinine ≤ 1.25x upper reference range

Exclusion Criteria:

* Previous radiotherapy, chemotherapy, surgery (excluding diagnostic biopsy) or any investigational drug for the NPC
* Concurrent chronic systemic immune therapy, targeted therapy, anti-VEGF therapy or EGFR-pathway targeting therapy not indicated in this study protocol
* Known hypersensitivity reaction to any of the components of study treatments
* Pregnancy or lactation period
* Systemic metastatic disease
* Clinically relevant coronary artery disease, history of myocardial infarction in the last 12 months, or high risk of uncontrolled arrhythmia
* Peripheral neuropathy > grade 1
* Previous malignancy except basal cell cancer of the skin or preinvasive cancer of the cervix
* Known alcohol or drug abuse
* Medical or psychological conditions that would not permit the patient to complete the study or sign informed consent
* Legal incapacity or limited legal capacity

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2010-05; Primary Completion 2013-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events as a measure of safety and tolerability | 1 year

SECONDARY OUTCOMES:
Objective response rate | 1 year
  Assess the response rate of this combination treatment, as measured by imaging and endoscopy findings
Progression and overall survival | 1 year
  To assess the PFS and OS at one year

CONTACTS AND LOCATIONS:
Overall Officials: Gwo Fuang Ho, FRCR, Principal Investigator — University of Malaya
Locations (1):
- University Malaya Medical Centre, Kuala Lumpur, Kuala Lumpur, Malaysia

DOCUMENTS (1):
  • Study Protocol (2019-01-04): https://cdn.clinicaltrials.gov/large-docs/76/NCT01230476/Prot_000.pdf